CLINICAL TRIAL: NCT04346082
Title: Feasibility and Acceptability of Online Based Mindfulness Interventions to Relieve Distress During COVID-19 Outbreak in a Chinese Population: a Proof-of-concept Trial
Brief Title: Feasibility of Online Based Mindfulness Interventions During COVID-19 Outbreak
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Regular mindfulness online sessions were not carried out
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: online-mind
Record Dates: First submitted 2020-04-07; First posted 2020-04-15 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Stress

STUDY DESIGN:
Intervention Model Description: participants receiving online mindfulness session(s)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- online mindfulness group (Experimental)
  Interventions: Behavioral: online mindfulness group

INTERVENTIONS:
Behavioral: online mindfulness group — Each weekly mindfulness session will last 45 to 60 minutes and will be held on an online platform (e.g. Zoom) via a livestream video. It will consist of short mindfulness exercise(s) of 10-30 minutes, including mindful tasting, mindful stretching, mindful walking, and body scan followed by group discussion to share, explore and make sense of the meditative experience. The intervention will be held in Cantonese.

SUMMARY:
The investigators had designed weekly mindfulness sessions (details see intervention below), which is free-of-charge and will be made available to general public who feel distressed during the outbreak of COVID-19. Face-to-face delivery of mindfulness interventions was not possible due to mandatory quarantine. The investigators hypothesize that this intervention is feasible and acceptable by the participants. As secondary outcomes, the investigators also hypothesize that the intervention can reduce stress, depressive and anxiety symptoms and enhance participants' sense of coherence

This will be a quasi-experimental study. Participants will be invited to fill in an online informed consent and questionnaire around 2 days before each mindfulness online session and another set of questionnaire immediately after each session (see outcome measures). Participants will be identified by their e-mail and therefore serial data could be obtained.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of old,
* able to speak and communicate in Cantonese
* can read Chinese or English (because they will be asked to fill in an online questionnaire).

Exclusion Criteria:

* actively suicidal,
* currently abusing restricted psychoactive substances
* diagnosed to have an active psychotic disorder and self-reported active psychotic symptoms (including schizophrenia, bipolar disorder and dementia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
rate of recruitment | from recruitment to end of study, up to 1 year
  the rate of recruitment to recruit participants
rate of attendence | from recruitment to end of study, up to 1 year
  the number of attendance to the mindfulness online group

SECONDARY OUTCOMES:
Depression, Anxiety and Stress Scale (DASS-21) | on recruitment, after each online mindfulness sessions (weekly) until end of study, up to 1 year
  Depression, anxiety and stress will be measured using the Depression, Anxiety and Stress Scale (DASS-21), which was validated in Chinese population with high internal consistency. The 21-item DASS-21 has three subscales designed to measure depression, anxiety and stress, with each subscale containing 7 items. Participants are required to rate each statement in DASS-21 using a 4-point Likert scale from "did not apply to me at all" to "applied to me very much or most of the time" in the prior one week. Higher scores represent higher level of psychological distress.
Sense of Coherence Scale | on recruitment, after each online mindfulness sessions (weekly) until end of study, up to 1 year
  Sense of Coherence (SOC) will be assessed by the 13-item Sense of Coherence Scale (SOC-13) based on Antonovsky (1987)'s measurement of the comprehensibility, manageability, and meaningfulness of a person's life events . Participants will rate each statement in SOC-13 on a 7-point Likert scale from "very often" to "very seldom or never". SOC-13 has been validated in Chinese population with high internal consistency. The higher the score, the higher the sense of coherence

CONTACTS AND LOCATIONS:
Locations (1):
- School of public health and primary care, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
may share data on request of investigators